CLINICAL TRIAL: NCT02208726
Title: The Effect of Picricum Acidum and Phosphoricum Acidum Homaccord on Perceived Levels of Anxiety in University Students
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr, University of Johannesburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KaronWillson200731900; AEC44-01-2013 (Other: University of Johannesburg)
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Anxiety
Keywords: anxiety; students; examinations; Homeopathy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sucrose pillules (Placebo Comparator): Unmedicated sucrose pillules will be taken once daily, in the morning, 30 minutes after breakfast, for 14 days, up to 7 days before the first academic examination.
  Interventions: Other: Sucrose pillules
- Homeopathic homaccord (Experimental): Sucrose pillules medicated with Picricum acidum and Phosphoricum acidum in potencies of 6CH, 30CH and 200CH. Pillules will be taken once daily, in the morning, 30 minutes after breakfast, for 14 days, up to 7 days before the first academic examination.
  Interventions: Other: Homeopathic homaccord

INTERVENTIONS:
Other: Sucrose pillules — Unmedicated sucrose pillules
  Other Names: Saccharum officinale
  Arms: Sucrose pillules
Other: Homeopathic homaccord — Sucrose pillules medicated with Picricum acidum and Phosphoricum acidum in potencies of 6CH, 30CH and 200CH.
  Other Names: Picricum acidum and Phosphoricum acidum homaccord
  Arms: Homeopathic homaccord

SUMMARY:
Increased levels of stress and anxiety are experienced by many students. Stress can have a negative influence on academic outcome and performance, as well as on the student's mental health. Conventional treatment options for anxiety include counseling, as well as anxiolytics and antidepressants, which may have various adverse effects. Picricum acidum and Phosphoricum acidum are homeopathic remedies that may be helpful in alleviating anxiety in students; however there has been no research done to date to show their efficacy for this condition.

The aim of this study is to determine the effect of Picricum acidum and Phosphoricum acidum Homaccord on perceived levels of anxiety in university students, by means of the State-Trait-Anxiety-Inventory and Anxiety Symptom Score Card.

DETAILED DESCRIPTION:
This study will be a randomized, double-blind, placebo-controlled study, conducted over a two-week period at the University of Johannesburg (UJ) Health Clinic, Doornfontein Campus. Thirty university students, aged between 18 and 45 years, will be recruited into the study by means of advertisements placed on the campus with relevant permission given. Participants will attend an initial consultation and will be requested to sign a Participant Information and Consent form, complete the Participant Information Sheet, and a Remedy Symptom Questionnaire to determine inclusion into the study. Participants' vital signs will be measured. Participants will then receive a 16ml vial of either the Picricum acidum and Phosphoricum acidum Homaccord pillules, or a placebo (unmedicated sucrose pillules), which will be randomized and dispensed by the UJ Homeopathic Dispenser. Participants will be requested to take 5 pillules in a daily dose for 14 days, commencing 21 days before and ceasing 7 days prior to the start of examinations. The State-Trait-Anxiety-Inventory (STAI) and the Anxiety Symptom Score Card will be completed 21 days prior to the first academic examination, as well as on the last day of taking the medication. Data will be collected and analyzed by Statkon, using the Shapiro-Wilk test, the Mann-Whitney test and the Wilcoxon signed ranks test.

The outcome of this research may show that the Homeopathic Picricum acidum and Phosphoricum acidum Homaccord has a positive effect in alleviating anxiety in university students, allowing for further studies in the field.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between the ages of 18 and 45;
* Registered University students;
* Participants must experience anxiety symptoms, manifesting six or more of the following criteria: muscle tension, increased perspiration, rapid heartbeat, headaches, stomach aches, agitation, irritability, hostility, fear, extreme sensitivity to rejection or failure, motor restlessness, procrastination, excessive worry, concentration difficulties, attention difficulties and memory problems;
* Participants must be writing a major examination one week after the study ends;
* Participants must have six or more of the symptoms relating to Picricum acidum and Phosphoricum acidum (Appendix D); and
* Participants must have a cell phone and on-line computer access.

Exclusion Criteria:

• Have been diagnosed with: A psychological anxiety disorder, Psychiatric disorders (Bipolar disorder, Depression), Attention Deficit Hyperactivity Disorder and Epilepsy.

* Are taking any chronic medication for anxiety or mood stabilizing
* Are pregnant or lactating

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
State-Trait-Anxiety-Inventory | 14 days
  The State-Trait-Anxiety-Inventory is an established, acceptably reliable, validated and commonly utilized tool for measuring an individual's level of anxiety.

SECONDARY OUTCOMES:
Anxiety Symptom Score Card | 14 days
  The Anxiety Symptom Score Card is based on a 5-point grading scale and is designed to monitor anxiety-related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Pellow, M.Tech Hom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No